CLINICAL TRIAL: NCT07061093
Title: Valutazione Prospettica Sul Ruolo Esercitato Dai Contraccettivi Ormonali Sulla Pressione Delle 24 Ore
Brief Title: Prospective Evaluation on the Role Exerted by Hormonal Contraceptives on 24-h Blood Pressure. A Prospective Observational Study
Acronym: HOLTER CO-PRE
Status: Recruiting | Type: Observational
Sponsor: Ospedale Policlinico San Martino (Other)
Responsible Party: Principal Investigator, Angelo Cagnacci, Full Professor Obstetric and Gynecology - Director Academic Unit of Obstetrics and Gynecology, Ospedale Policlinico San Martino
Other Study IDs: 12674
Record Dates: First submitted 2025-07-02; First posted 2025-07-11 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Cardiovascular System Diseases (&Amp; [Cardiac])
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Ethinyl Estradiol; drospirenone; drospirenone and estetrol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Ethynyl estradiol and Drospirenone — Oral ethynyl estradiol (20 mcg) and 3 mg drospirenone for 24 days and 4 days free of hormones
Drug: Drospirenone — A drospirenone (4mg) only pill
Drug: Estetrol and Drospirenone — Oral estetrol (15 mg) and drospirenone (3 mg) for 24 days and 4 days of interval free of hormone

SUMMARY:
This study aims to assess the effect of different hormonal contraceptives on 24-h blood pressure in cycling women aged 18-50 years of age.

The main question aims to answer:

- Does oral contraceptives, estrogen formulations' based combined with drospirenone or the only drospirenone present minr effect on blod pressure and/or on the heart rate?

Participants will:

* Receive a contraceptive for at least 4 months
* Visit the clinic between days 3 and 8 of the menstrual cycle for recording of vital signs and 40 hours-blood pressure monitoring every 30 min from 17.00 to 8.00 of the following second day
* Have a gynecological examination performed at screening and at cycle 4

DETAILED DESCRIPTION:
Aim of this study is to investigate a possible minor effect on blood pressure and, secondarily, on heart rate of oral contraceptives based on the new estrogen formulations combined with drospirenone or with the administration of drospirenone alone.

The seecondary objectives are:

* To evaluate modification of prevalence of dippers and non-dippers for each treatment
* To evaluate 24-h variation of Heart Rate For all women participating in this trial the total treatment period is at least 4 consecutive cycles of 28 days each.

The experimental flow will have a:

* Screening phase: inform the subject, orally and in writing, about the purpose, procedures, and general risks of participating in the trial and collect all data required
* Baseline phase: the investigation is performed in the follicular phase between days 3 and 8 of the menstrual cycle; recording of height, body weight and blood pressure, and an ulterior 40 hours-blood pressure monitoring -Cycle 4 phase: in which the recording made during the Baseline phase will be repeated-

ELIGIBILITY:
Inclusion Criteria:

* Sexually active women, at risk for pregnancy and willing to use a contraceptive for at least 4 cycles
* Women with regular menstrual cycles with an intermenstrul period between 21 and 35 days
* An age between 18 and 50 years at time of screening
* Body mass index ≥18 and ≤30;
* Good physical and mental health;
* Choose either no hormonal contraception or one of the specific contraceptives under investigation
* Willing to give informed consent in writing

Exclusion Criteria:

* Contraindications for contraceptive steroids:

  * Presence or a history of venous or arterial thrombotic/thromboembolic events (e.g. deep venous thrombosis, pulmonary embolism, myocardial infarction) or of a cerebrovascular accident;
  * Precence or history of prodromi of a thrombosis (e.g. transient ischaemic attack, angina pectoris);
  * History of migraine with focal neurological symptoms;
  * Diabetes mellitus with vascular involvement;
  * The presence of a severe or multiple risck factor(s) for venous or arterial thrombosis (to be judged by the (sub)-investigator).

    e.g. increasing age; smoking (with heavier smoking and increasing age the risk further increases, especially in women over 35 years of age); a positive family history (i.e. venous or arterial thromboembolism ever in a sibling or parent at an age< 40 years o); obesity (body mass index over 30 kg/m2); dyslipoproteinaemia; hypertension, migraine, valvular heart disease, atrial fibrillation; prolonged immobilization, major surgery any surgery to the legs, or major trauma (until two weeks after full remobilization); systemic lupus erythematosus; haemolytic uraemic syndrome; chronic inflammatory bowel disease (Crohn's disease or ulcerative colitis); sickle cell disease;
  * Severe dyslipoproteinemia
  * Blood pressure above 140/90 mmHg
  * Known hereditary or acquired predisposition for venous or arterial thrombosis, such as APC resistance, antithrombin-lll-deficiency, protein C deficiency, protein S deficiency, hyperhomocysteinaemia and antiphospholipid antibodies (anticardiolipin antibodies, lupus anticoagulant);
  * Pancreatitis or a history thereof if associated with severe hypertriglyceridaemia;
  * Presence or history of severe hepatic disease as long as liver function values have not returned to normal;
  * Presence or history of liver tumors (benign or malignant);
  * Known or suspected sex steroid-influenced malignancies (e.g. of the genital organs or the breasts);
  * Undiagnosed vaginal bleeding
  * Known or suspected pregnancy
  * Hypersensitivity to the active substances or to any of the excipients of the investigational product
* An abnormal cervical smear (i.e.: dysplasia, cervical intraepithelial neoplasia (CIN), SIL, carcinoma in situ, invasive carcinoma) at the screening evaluation
* Clinically relevant abnormal laboratory data as judged by the investigator;
* Post-partum (6 months from delivery)
* Breastfeeding or 2 months from breastfeeding ending
* Present use or use in the last 2 months of the following drugs: phenytoin, barbiturates, primidone, carbamazapine, oxcarbazepine, topiramate, felbamate, rifampicin, nelfinavir, ritonavir, griseofulvin, ketoconazole, sex steroids (other than pre- and post-treatment contraceptive method) and herbal remedies containing Hipericum perforatum (St John's Wort);
* Administration of any other investigational drugs and/or participation in other clinical trial in the last 2 months.
* Present use of any oral contraceptive.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Subjects will be recruited from outpatient hospital centre for contraception at the University Hospital San Martino of Genova (Italy). Subjects can only be included in the trial if all inclusion criteria are fulfilled, while none of the exclusion criteria are present.
Sampling Method: Probability Sample
Enrollment: 96 (Estimated)
Dates: Start 2023-10-10 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Rhythmometric evaluation by cosinor analysis | From starting of the treatment to the end of it at 4 months
  When cosinor analysis is significant, we calculate and record the nadir (time of minimal cosine function; that is, the time in the 24-h period when mean BP and heart rate are at their theoretical minimum). Rhythms are put in phase by considering the nadir as the circadian time 0. The 24-h, daytime, and night-time (3 h before and 3 h after the time of nadir) values are separately evaluated. Assuming a difference in blood pressure o heart rate of 3 mmHg with a standard deviation of the difference of 6 mmHg and setting type I error at 0.05 and type II error at 0.20, 32 women need to be enrolled in each group of treatment.

SECONDARY OUTCOMES:
Comparison of modifications induced by treatments | From starting of the treatment to the end of it at 4 months
Identification of the parameters conditioning the eventual BP or heart rate response to treatments | From starting of the treatment to the end of it at 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Angelo Cagnacci, MD, PhD, Principal Investigator — Clinica Ostetrica e Ginecologica, IRCCS-Ospedale San Martino di Genova
Locations (1):
- Ospedale San Martino, Genova, GE, Italy